CLINICAL TRIAL: NCT01524627
Title: Characterizing a Cue-vulnerable Pharmaco-responsive Endophenotype in Smokers
Brief Title: Effects of Varenicline on Smoking Reminders
Acronym: VSMK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 813779; 1R01DA029845-01A1 (NIH)
Record Dates: First submitted 2012-01-10; First posted 2012-02-02 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Nicotine Dependence
Keywords: Smokers; fMRI; varenicline
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): Placebo will be prescribed to non-abstinent smokers at the same doses as have been demonstrated to be clinically effective for Varenicline: 0.5 mg twice a day for 3 days and then 1mg twice daily for the remainder of the treatment course of 8 weeks.
  Interventions: Drug: Placebo
- Varenicline (Active Comparator): Varenicline will be prescribed to non-abstinent smokers at the same doses as have been demonstrated to be clinically effective: 0.5 mg twice a day for 3 days and then 1mg twice daily for the remainder of the treatment course of 8 weeks.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline will be prescribed to non-abstinent smokers at the same doses as have been demonstrated to be clinically effective: 0.5 mg twice a day for 3 days and then 1mg twice daily for the remainder of the treatment course of 8 weeks.
  Other Names: Chantix
  Arms: Varenicline
Drug: Placebo — Placebo will be prescribed to non-abstinent smokers at the same doses as have been demonstrated to be clinically effective for Varenicline: 0.5 mg twice a day for 3 days and then 1mg twice daily for the remainder of the treatment course of 8 weeks.
  Other Names: Sugar Pill
  Arms: Control Group

SUMMARY:
Varenicline is the best smoking cessation agent to date; however it is only effective in a subgroup of smokers and is associated with undesirable side effects in other subgroups. To understand the underlying pharmaco-heterogeneity, the proposed project will use perfusion functional magnetic resonance imaging and a functional candidate gene association approach using brain, behavioral, and clinical endpoints in a placebo-controlled study of chronic varenicline administration in smokers. Brain and behavioral responses to smoking cues will be will be significantly greater in 9/10-repeats compared to 10/10-repeats. DAT 9/10-repeat smokers receiving varenicline will have better treatment outcome compared to 10/10-repeats. For the purposes of the clinical trial portion of the study, the change from cigarettes per day at Baseline to the last day of treatment will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy male or female nicotine dependent patients ages 18-60 without other current drug dependence or psychiatric diagnosis.
* Smoke ≥ 10 cigarettes per day for at least 6 months prior to study start date.
* Females must be non-pregnant, non-lactating and either be of non-childbearing potential (i.e. sterilized via hysterectomy or bilateral tubal ligation or at least 1 year post-menopausal) or of child bearing potential but practicing a medically acceptable method of birth control from at least 2 weeks prior to screening until 30 days after the last dose of varenicline. Examples of medically acceptable methods for this protocol include barrier (diaphragm or condom) with spermicide, an intrauterine (IUD), oral contraceptives, levonorgestrel implant, or complete abstinence.
* Subjects provide voluntary informed consent.
* Subjects must read at 8th grade level or higher.

Exclusion Criteria:

* History of head trauma or injury causing loss of consciousness, lasting more than three (3) minutes or associated with skull fracture or inter-cranial bleeding or abnormal MRI.
* Presence of magnetically active prosthetics, plates, pins, permanent retainer, bullets, etc. in patient's body (unless a radiologist confirms that it's presence is unproblematic). An x-ray may be obtained to determine eligibility given the possibility of a foreign body.
* Self report of HIV positive and on medication for symptoms: Determined on an individual basis by results from the physical examination and final approval by the study physician.
* Symptomatic presence of other hematological disease.
* Clinically significant hepatic (liver), renal (kidney), neurological, or endocrinological abnormalities.
* History of any cardiovascular event within the last 6 months and any serious/significant cardiovascular event in the subject's life. This will be determined on an individual basis by the study physician.
* History of psychosis or seizures.
* Use of medications or natural herbs that may cause sedation or may effect the brain systems that are being studied (medication use will be evaluated on a case-by-case basis).
* Claustrophobia or other medical condition preventing subject from lying in the MRI for approximately one (1) hour.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2011-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Franklin, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Addiction Treatment Research Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1/2012-7/2015. Methods used to recruit were flyers, advertisements on public transportation, Craigslist, word of mouth.
  596 potential subjects were phone screened, 124 of those successfully consented, 43 were randomized
Groups:
- Placebo: Placebo will be prescribed to non-abstinent smokers at the same doses as have been demonstrated to be clinically effective as Varenicline: 0.5 mg twice a day for 3 days and then 1mg twice daily for the remainder of the treatment course of 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Varenicline
Started | 22 | 21
Completed | 21 | 19
Not Completed | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants will receive either varenicline or placebo
  Varenicline or placebo: Varenicline or placebo will be prescribed to non-abstinent smokers at the same doses as have been demonstrated to be clinically effective: 0.5 mg twice a day for 3 days and then 1mg twice daily for the remainder of the treatment course of 8 weeks.
- Varenicline: Subjects will receive either varenicline or placebo
  Varenicline or placebo: Varenicline or placebo will be prescribed to non-abstinent smokers at the same doses as have been demonstrated to be clinically effective: 0.5 mg twice a day for 3 days and then 1mg twice daily for the remainder of the treatment course of 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Varenicline | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (11.1) | 36.2 (11.9) | 38.1 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 11 | 9 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 12 | 18
  Black | 15 | 8 | 23
  Asian | 1 | 0 | 1
  Mixed Race | 0 | 1 | 1
  Hispanic | 3 | 1 | 4
  Non-Hispanic | 18 | 21 | 39
Region of Enrollment [Number; unit: participants]
  United States | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Cigarettes Per Day
Description: Cigarettes per day at Baseline versus 8 weeks of treatment, placebo-controlled
Time Frame: last week of treatment (1-8 weeks)
Population: Population was the number of randomized subjects who participated in any treatment length. One subject per group was not included in this analysis as one withdrew a few days after their first scan and the other was lost to follow up after their first scan.
Measure: Mean (Standard Error); unit: cigarettes per day
Arm/Group | Placebo | Varenicline
Number analyzed (Participants) | 21 | 20
cigarettes per day
  Baseline | 15.7 (2.5) | 14.3 (1.8)
  Following Treatment | 9.8 (2.6) | 5.3 (1.6)
Statistical Analysis 1: Comparison: Varenicline; Test type: Superiority; p = 0.0004, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo; Test type: Superiority; p = 0.1, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Collected over 5 years during a subject's week 1-8
Arm/Group | Placebo | Varenicline
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 13/22 | 8/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | Varenicline (N=21)
Coughing (mild) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dizziness (mild) (Nervous system disorders) | 3 (3) | 0 (0)
Headache (mild) (Nervous system disorders) | 5 (5) | 0 (0)
Nausea (mild) (Gastrointestinal disorders) | 3 (3) | 7 (10)
Nausea (moderate) (Gastrointestinal disorders) | 2 (2) | 2 (2)
Sedation/Drowsiness (mild) (Nervous system disorders) | 3 (3) | 2 (2)
Skin Irritation (mild) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Vivid Dreams (mild) (Nervous system disorders) | 2 (5) | 0 (0)
Upper Respiratory Infection (moderate) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes